CLINICAL TRIAL: NCT06345092
Title: Comparison Between Injectable Platelet Rich Fibrin With Vitamin C and Injectable Platelet Rich Fibrin Alone in Management of ID'Pain
Brief Title: Comparison Between IPRF With Vit. C and IPRF Alone in Management of ID'Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youmna alaa yehia, MSc degree of oral and maxillofacial surgery Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omfs.3-3-3
Record Dates: First submitted 2024-03-26; First posted 2024-04-03 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: TMJ Pain
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): injection of injectable platelet rich fibrin with vitamin C
  Interventions: Drug: Vitamin C; Other: Injectable platelet rich fibrin
- control group (Active Comparator): injection of injectable platelet rich fibrin alone
  Interventions: Other: Injectable platelet rich fibrin

INTERVENTIONS:
Drug: Vitamin C — addition of vitamin C to IPRF
  Other Names: Ascorbic acid
  Arms: intervention group
Other: Injectable platelet rich fibrin — injection of IPRF alone
  Other Names: IPRF

SUMMARY:
Randomized clinical trial between 2groups,the study group to be injected in the TMJ with injectable platelet rich fibrin with vitamin C and the control group to be injected in the TMJ with injectable platelet rich fibrin alone in management of internal Temporomandibular joint derangement

DETAILED DESCRIPTION:
Randomized clinical trial between 2groups,the study group to be injected in the TMJ with injectable platelet rich fibrin with vitamin C and the control group to be injected in the TMJ with injectable platelet rich fibrin alone in management of internal Temporomandibular joint derangement

ELIGIBILITY:
Inclusion Criteria:

Patients with internal TMJ derangement (anterior disc displacement with reduction)

Exclusion Criteria:

Pathological conditions ; trauma TMJ cases or any blood diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pain management | at 4;8;12;16 weeks
  Evaluation of pain using VAS pre and post injections

SECONDARY OUTCOMES:
disc position using MRI | at 4;8;12;16 weeks
  evaluation of disc position pre and post injections

OTHER OUTCOMES:
maximum mouth opening | at 4;8;12;16 weeks
  measurement of MMO using digital caliper pre and post injections
lateral excursion | at 4;8;12;16 weeks
  measurement of lateral excursion using digital caliper pre and post injections

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry cairo university, Cairo, Egypt